CLINICAL TRIAL: NCT04349982
Title: Prospective Observational ICU Trial in Critical Ill COVID-19 Patients (POINT-C) Cardiovascular Risk and the Effects on Myocardial Events in Critical Ill COVID-19 Patients
Brief Title: ICU Trial in Critical Ill COVID-19 Patients
Acronym: POINT-C
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Martin Rief, Dr., Medical University of Graz
Other Study IDs: 250320
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Risk Factor, Cardiovascular; Covid19; Critical Illness; Course Illness
Keywords: Critical Illness; Covid19; Risk Factor, Cardiovascular
MeSH Terms: conditions — COVID-19; Critical Illness; Disease Progression | interventions — Prone Position; Inhalation; Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Lipid profile once at intensive care unit admission (9 ml whole blood).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No cardiovascular risk: If no patients with no cardiovascular risk can be included in the study, we will divide the cohorts into different categories (e.g. low, medium and high cardiovascular risk).
  Interventions: Diagnostic Test: Biomarker (TropT, Myoglobin, CK, CK-MB, LDH, D-dimer, CRP, PCT)
- low cardiovascular risk
  Interventions: Diagnostic Test: Biomarker (TropT, Myoglobin, CK, CK-MB, LDH, D-dimer, CRP, PCT)
- high cardiovascular risk
  Interventions: Diagnostic Test: Biomarker (TropT, Myoglobin, CK, CK-MB, LDH, D-dimer, CRP, PCT)

INTERVENTIONS:
Diagnostic Test: Biomarker (TropT, Myoglobin, CK, CK-MB, LDH, D-dimer, CRP, PCT) — Factorial
  Other Names: Fluid management (fluid input, fluid output), prone positioning, ventilation, respiration, circulation parameters, extracorporeal organ support procedures, mortality, MACE, entire drug therapy

SUMMARY:
The aim of our study is to observe the intensive care course in 30-50 COVID-19 patients with regard to cardiovascular risk factors and biomarkers.

The primary objective of this study is to investigate the cardiovascular risk and its impact on cardiovascular complications in COVID-19 patients in intensive care units.

This study is designed to investigate correlations and to investigate factors influencing the course of the new viral disease COVID-19 in intensive care. Previous scientific findings are still rare due to the relevance of the disease, therefore this study is also explorative and not exclusively based on a hypothesis.

The cardiovascular risk will be assessed upon admission to the intensive care unit and subsequently the course of biomarkers (see below) will be analysed in a cohort study (no, low and high cardiovascular risk).

DETAILED DESCRIPTION:
In this prospective observational study the course of 30-50 intensive care patients of the University Hospital of Graz is analysed.

It is not possible to give an exact number of cases, because it is not possible to estimate exactly how many COVID-19 patients will be admitted to the listed intensive care units in Graz. Recruitment will start when approved from the ethical board and end in June, 2020.

Inclusion criteria

* Admission on an isolation unit - intensive care unit of the University Clinic of Graz
* Detection of a SARS - CoV-2 infection by PCR (tracheal or pharyngeal secretion) or CT examination (with consecutive PCR confirmation)
* male and female sex
* subordinated declaration of consent if possible*
* respiratory insufficiency with indication for non-invasive or invasive ventilation during admission to an intensive care unit

Informed consent

Since the study patients are intensive care patients, it may happen that the informed consent cannot be obtained at the time of admission to the intensive care unit (e.g.: patient is not able to give consent due to mechanical ventilation), in this case the informed consent will be obtained at a later time (e.g.: at the latest upon discharge from the intensive care unit/hospital.

(* In exceptional cases it may happen that patients cannot sign a declaration of consent at admission as well as at discharge from the intensive care unit (e.g.: during the stay continuous mechanical ventilation and death at the intensive care unit).

Study related measures

In addition to the standardized routine laboratory (daily, in the morning approx. 05.00 o'clock), a lipid profile (LDL cholesterol, triglycerides, Lpa, HDL cholesterol, total cholesterol) is taken once upon admission to the intensive care unit in order to determine the cardiovascular risk upon admission to the intensive care unit. This lipid profile is taken with the aid of a vacuette (9 ml corresponds to approx. 2 teaspoons of whole blood).

Study related patient questionnaire for the determination of cardiovascular risk

The patient questionnaire should be filled out by interviewing the patients at the time of admission to the intensive care unit. If the condition of the patients does not allow this, the information in the questionnaire should be carried out by a member of the study staff by researching the patient's medical history (e.g. doctor's letters, electronic data acquisition, etc.). The questionnaire is used to assess the cardiovascular risk (contains medication, past medical history).

Non-study-related measures (standardised routine analyses in an intensive care unit)

To determine the cardiovascular risk:

See Patient Questionnaire, Lipid Status, HbA1c

For follow-up (daily routine laboratory checks):

Blood count, coagulation, liver and kidney counts, triglycerides, biomarkers (CK, CK-MB, TropT, NTproBNP, CRP, PCT, IL-6, D-dimer, LDH, myoglobin).

Other parameters and therapies that are considered in the evaluation or that are used to create the data set:

Fluid introduction, fluid discharge, balance, prone positioning, non-invasive ventilation (PEEP, fiO2), invasive ventilation (ventilation mode, PEEP, Pinsp, fiO2, AF), respiration (respiratory rate, fiO2, SpO2, paO2, pCO2, etCO2), circulation parameters (RR syst, RR dia, MAP, HF, ECG (rhythm, Qtc)), extracorporeal organ support procedures, mortality, med. complications, entire drug therapy (e.g: norepinephrine (incl. dose), levosimendan (incl. dose), vasopressin (incl. dose), cortisone (incl. dose), dobutamine (incl. dose), supportive therapy (zinc, vitamin C, selenium), antifungal and antibiotic therapy, hydroxychloroquine, lopinavir, remdesivir, favipiravir, tocilizumab.

Anonymisation of patients

After enrolment in the study, the patient data is encoded/pseudo-anonymised, i.e. patients are identified with a consecutive ID number (neither name, initials nor laboratory requirement number are recorded). To find out the previous illnesses of intensive care patients it is necessary to create a list of patient names and the corresponding ID numbers for pseudonymisation. This list remains with the investigator.

Use of clinical data For the statistical analysis, clinical data in pseudo-anonymised/encoded form are used, e.g. diagnosis, concomitant diseases, long-term medication, intensive care therapy, medication, smoking, age, sex.

Should further questions arise during the study regarding this patient collective, the collected data would be used for further evaluations.

Centre/intensive care units The test centre is the LKH Univ.Klinikum Graz, Auenbruggerplatz 5, A-8036 Graz. Patients are admitted to the SARS - CoV-2 (COVID-19) isolation unit intensive care units of the LKH University Hospital Graz.

ELIGIBILITY:
Inclusion Criteria:

* Admission on an isolation unit - intensive care unit of the LKH Univ. Klinikum Graz
* Detection of a SARS - CoV-2 infection by PCR (tracheal or pharyngeal secretion) or CT examination (with subsequent PCR detection)
* male and female sex
* subordinated declaration of consent if possible if applicable
* respiratory insufficiency with indication for non-invasive or invasive ventilation

Exclusion Criteria:

* if the inclusion criteria are not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respiratory insufficiency and current COVID-19 infection with different gender, age and previous diseases.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
ICU CV risk and Biomarker (e.g. Troponin) | through study completion, up to 4 weeks
  Troponin courses in the intensive care unit are analyzed in consideration of the respective cardiovascular risk.

SECONDARY OUTCOMES:
CV risk and Outcome during ICU stay | through study completion, up to 4 weeks
  The 30-day mortality during the ICU stay is determined and divided into appropriate cardiovascular risk groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
If other researchers need the medical data of this study for their research projects, the data will be made available after consideration for co-autorship.

REFERENCES:
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Li B, Yang J, Zhao F, Zhi L, Wang X, Liu L, Bi Z, Zhao Y. Prevalence and impact of cardiovascular metabolic diseases on COVID-19 in China. Clin Res Cardiol. 2020 May;109(5):531-538. doi: 10.1007/s00392-020-01626-9. Epub 2020 Mar 11. PMID 32161990
- [Background] Lippi G, Lavie CJ, Sanchis-Gomar F. Cardiac troponin I in patients with coronavirus disease 2019 (COVID-19): Evidence from a meta-analysis. Prog Cardiovasc Dis. 2020 May-Jun;63(3):390-391. doi: 10.1016/j.pcad.2020.03.001. Epub 2020 Mar 10. No abstract available. PMID 32169400
- [Background] Yang J, Zheng Y, Gou X, Pu K, Chen Z, Guo Q, Ji R, Wang H, Wang Y, Zhou Y. Prevalence of comorbidities and its effects in patients infected with SARS-CoV-2: a systematic review and meta-analysis. Int J Infect Dis. 2020 May;94:91-95. doi: 10.1016/j.ijid.2020.03.017. Epub 2020 Mar 12. PMID 32173574